CLINICAL TRIAL: NCT01437709
Title: Ofatumumab With or Without Bendamustine for Patients With Mantle Cell Lymphoma Ineligible for Autologous Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-050
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: Bendamustine HCL; Ofatumumab (GSK 1841157); Immunotherapy; Chemoimmunotherapy; 11-050
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ofatumumab; Bendamustine Hydrochloride

ARMS (2):
- patients receiving Immunotherapy (This arm is closed) (Experimental): The proposed study is a Simon 2 stage optimal study design investigating the activity of ofatumumab alone or in conjunction with Bendamustine for patients with MCL who are either not candidates for ASCT or aged 65 or older. The study design will allow for an estimation of the single agent response of ofatumumab in patients at low biologic risk for immediate disease progression.
  Interventions: Biological: Ofatumumab (This arm is closed)
- patients receiving Chemoimmunotherapy (Experimental): The proposed study is a Simon 2 stage optimal study design investigating the activity of ofatumumab alone or in conjunction with Bendamustine for patients with MCL who are either not candidates for ASCT or aged 65 or older. The combined regimen will assess the response rates of the combined chemo- immunotherapy program in patients with need for cytoreductive therapy, or high risk for disease progression. Patients with a leukemic phase only presentation of mantle cell lymphoma generally have clinically low-risk disease, regardless of mantle cell IPI calculations. Upon reciew with the principal investigator, these patients may be stratified to the immunotherapy only arm if clinically appropriate.
  Interventions: Other: Ofatumumab + Bendamustine

INTERVENTIONS:
Biological: Ofatumumab (This arm is closed) — Ofatumumab Day 1 Week 1: 1000 mg, Day 2 week 1: 1000mg. Patients who exhibit a baseline leukocytosis ≥ 20,000 will receive 300 mg of ofatumumab on day 1, week 1. Thereafter, they can receive the 1000 mg dose Ofatumumab Day 1, Weeks 2-4: 1000 mg Will reassess 8-10 weeks after conclusion of treatment with CT CAP, and following this q 12 wks for 2 yrs, then q 6mo until POD or for a maximum of 5 years
  Arms: patients receiving Immunotherapy (This arm is closed)
Other: Ofatumumab + Bendamustine — Ofatumumab day 1 + Bendamustine 90 mg/m2 days 1 & 2 x 6 cycles q 28 days Cycle 1, day 1: Ofatumumab 1000 mg followed by Bendamustine 90 mg/m2. Patients who exhibit a leukocytosis ≥ 20,000 will receive 300 mg of ofatumumab on day 1, week 1. Thereafter, they can receive the 1000 mg dose. Cycle 1, day 2: Ofatumumab 1000mg followed by Bendamustine 90 mg/m2 Cycles 2-6: Ofatumumab 1000 mg day 1, Bendamustine 90 mg/m2 days 1 and 2 Will reassess 4-6 weeks after conclusion of treatment with CT CAP, and following this q 12 wks for 2 yrs, then q 6mo until POD or for a maximum of 5 years
  Arms: patients receiving Chemoimmunotherapy

SUMMARY:
This study is being done to understand how to treat Mantle Cell Lymphoma (MCL). The goals of treatment are to control the lymphoma with the least amount of side effects. In many cases, MCL is treated with an antibody plus chemotherapy. An antibody is a laboratory-produced substance created to attach to proteins on the cancer cells, eventually destroying them. Chemotherapy is medicine that specifically destroys cancer cells.

The purpose of this study is to find out what effects, good and/or bad, the drugs Ofatumumab and Bendamustine have on this type of cancer. Patients in this study will either receive Ofatumumab alone, or Ofatumumab combined with Bendamustine.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, non-transplant eligible, newly diagnosed mantle cell lymphoma with measurable disease as determined by CT, and bone marrow biopsy.
* Age > or = to 65 years or > 18 year and ineligible for HDT/ASCT.
* Subjects must not be candidates for intensive high-dose chemotherapy, with or without an autologous stem cell transplant (ASCT), due to one or more of the following factors:
* Age ≥ 65 years
* Patients <65 years of age must be ineligible for HDT/ASCT on the basis of comorbidity, organ dysfunction or patient refusal for HDT/ASCT Comorbid disease, such as CAD, CHF, pulmonary dysfunction, liver or kidney dysfunction, precluding high dose therapy secondary to expected increased morbidity and mortality.
* poor performance status (KPS 70% or less)
* Ejection fraction <45%
* Impaired pulmonary function test with DLCO <50% expected
* Patient refusal
* Medical conditions which in the opinion of the treating physician and DMT preclude HDT/ASCT.
* Patients must have a serum creatinine clearance ≥ 40 mL/min (as per the Jelliffe method) or by 12-hour or 24-hour urine creatinine clearance.
* Patients must have ANC>1,000/mcl and Platelets>100,000/mcl (unless secondary to MCL).
* Patients must have a bilirubin level of < 2.0 mg/dl in the absence of a history of Gilbert's disease (or pattern consistent with Gilbert's).
* Negative serologies for Hepatitis B (HB) defined as a negative test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if negative, patient may be included but must undergo HBV DNA PCR testing at the beginning of treatment and throughout treatment duration, at least every 2 months. In addition patients will require treatment with Entacavir .5mg po qday per MSKCC institutional guidelines.
* No active co-morbid cardiac condition such as active CHF or CAD.
* KPS performance ≥ 70%.
* Histologically confirmed mantle cell lymphoma classified according to WHO criteria confirmed at MSKCC.
* No prior treatment for mantle cell lymphoma with the exception of corticosteroids for 7 days or less or 1 course of involved-field radiation.
* No prior malignancies within 5 yrs, unless treated early stage breast cancer, treated carcinoma in situ of the cervix, resected skin malignancies, or treated prostate cancer.
* Women who are pre-menopausal must have a negative serum pregnancy test. Subjects must agree to use appropriate contraception until 4 weeks after the completion of chemotherapy.
* Patients must be HIV negative, and have negative serologies for Hepatitis C.

Exclusion Criteria:

* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, hepatic involvement by MCL, or stable chronic liver disease per investigator assessment).
* Known pregnancy or breast-feeding.
* Medical illness unrelated to MCL within the prior one month that will preclude administration of chemotherapy safely. This includes patients with uncontrolled infection, chronic renal insufficiency, myocardial infarction within the past 6 months, unstable angina, active congestive heart failure, cardiac arrhythmias other than chronic atrial fibrillation and chronic active or persistent hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hamlin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab: Ofatumumab alone for patients with MCL who are either not candidates for ASCT or aged 65 or older.
- Ofatumumab + Bendamustine: Ofatumumab + Bendamustine for patients with MCL who are either not candidates for ASCT or aged 65 or older.
- Ofatumumab Progressors: Ofatumumab alone participants who progressed and then received Ofatumumab + Bendamustine
Period: Overall Study
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
Started | 3 | 24 | 3
Completed | 3 | 22 | 3
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Pt trasnferred care | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors | Total
Number analyzed (Participants) | 3 | 24 | 3 | 30
Age, Continuous [Median (Full Range); unit: years] | 55 [46 to 75] | 73 [44 to 89] | 71 [68 to 73] | 73 [44 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 1 | 5
  Male | 3 | 20 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 20 | 3 | 26
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 18 | 3 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 24 | 3 | 30

OUTCOME MEASURES:

1. Primary Outcome: Single Agent Efficacy (as Determined by Response Rate)
Description: of the monoclonal antibody ofatumumab alone in low risk patients. Assessments prior to each cycle of immunotherapy or chemoimmunotherapy: (every 4 weeks)
Time Frame: 2 years
Population: Dual therapy arm not assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
Number analyzed (Participants) | 3 | 0 | 0
Participants
  Complete Response | 1 |  |
  No Response | 2 |  |

2. Primary Outcome: the Efficacy (as Determined by Response Rate) of the Combination Ofatumumab + Bendamustine
Description: in high risk patients. Assessments prior to each cycle of immunotherapy or chemoimmunotherapy: (every 4 weeks)
Time Frame: 2 years
Population: Single therapy arm not assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
Number analyzed (Participants) | 0 | 24 | 3
Participants
  Complete Response |  | 16 | 2
  No Response |  | 8 | 1

3. Secondary Outcome: Overall Survival (OS)
Description: will be analyzed using Kaplan-Meier estimation, and logrank tests or Cox regression models when covariates are involved.
Time Frame: Up to 6 years
Population: Participants in Ofatumab Progressors group were included in overall survival calculations for both ofatumumab single-agent and ofatumumab + bendamustine chemotherapy groups because this group consists of participants who were originally assigned to the single treatment arm who then progressed and then received dual therapy treatment.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
Number analyzed (Participants) | 3 | 24 | 0
years | 2.2 [0.25 to 4.8] | 5.8 [5.8 to NA] — Not Reached |

4. Secondary Outcome: Progression Free Survival (PFS)
Description: will be analyzed using Kaplan-Meier estimation, and logrank tests or Cox regression models when covariates are involved.
Time Frame: 2 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
Number analyzed (Participants) | 3 | 24 | 0
years | 0.31 [0.28 to NA] — Not Reached | 2.0 [1.5 to 4.8] |

5. Secondary Outcome: Remission Duration
Description: (calculated from confirmation of CR to progression)will be analyzed using competing risks tools (with death as a competing risk for progression), and will be done on the subsets of patients who have CR or CR/PR.
Time Frame: Up to 6 years
Population: Only participants considered responders were assessed
Measure: Median (Full Range); unit: years
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
Number analyzed (Participants) | 1 | 16 | 2
years | 3.36 [NA to NA] — Only 1 participant fulfilled the criteria for outcome measure 5 | 1.46 [0.11 to 5.66] | 2.45 [1.91 to 2.98]

6. Secondary Outcome: Response Duration
Description: (calculated from confirmation of response (CR/PR) to progression. will be analyzed using competing risks tools (with death as a competing risk for progression), and will be done on the subsets of patients who have CR or CR/PR.
Time Frame: Up to 6 years
Population: Only participants considered responders were assessed.
Measure: Median (Full Range); unit: years
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
Number analyzed (Participants) | 1 | 16 | 2
years | 4.19 [NA to NA] — Only 1 participant fulfilled the criteria for outcome measure 6 | 1.67 [0.36 to 5.93] | 2.79 [2.20 to 3.37]

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Ofatumumab | Ofatumumab + Bendamustine | Ofatumumab Progressors
All-Cause Mortality (participants affected / at risk) | 1/3 | 13/24 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 7/24 | 1/3
Other Adverse Events (participants affected / at risk) | 1/3 | 23/24 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=3) | Ofatumumab + Bendamustine (N=24) | Ofatumumab Progressors (N=3)
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 0
Infection, NOS (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Malignant neoplasm, NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=3) | Ofatumumab + Bendamustine (N=24) | Ofatumumab Progressors (N=3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 11 | 1
Fatigue (General disorders) | 0 | 10 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 10 | 3
Lymphocyte count decreased (Investigations) | 0 | 10 | 1
White blood cell decreased (Investigations) | 0 | 10 | 0
Neutrophil count decreased (Investigations) | 0 | 6 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 5 | 0
Fever (General disorders) | 0 | 5 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0
Blurred vision (Eye disorders) | 0 | 2 | 0
Chills (General disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 2 | 0
Edema limbs (General disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT01437709/Prot_SAP_000.pdf